CLINICAL TRIAL: NCT07344493
Title: Average ANKLE GO Score in the Objective Functional Assessment of the Ankle in Healthy Military Personnel (ANKMIL)
Acronym: ANKMIL
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2025PPRC07
Record Dates: First submitted 2025-11-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ankle Disorders Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to establish reference values for the Ankle-Go score, a validated tool for functional assessment of the ankle, in healthy military personnel. The Ankle-Go score, already used in the civilian population after sprains or surgery, combines physical tests and subjective questionnaires to assess functional recovery of the ankle. No normative data currently exist for the military population, whose physical and operational requirements differ significantly from those of the general population. This is an observational, prospective, single-center study conducted at the 39th medical branch in Oberhoffen (5th CMA). It will include 96 active military personnel with healthy ankles, examined during their periodic medical visit. Participants will complete the full Ankle-Go test and fill out the associated questionnaires on the secure anklego.com platform. The data will then be analyzed anonymously to calculate a reference average and explore possible variations according to gender and age. These results will ultimately improve care and fitness-to-duty decisions after ankle injuries in the military. The total duration of the study is estimated at 8 months, including 6 months of data collection and 2 months of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Active military personnel assigned to the 39th Medical Unit in Oberhoffen (5th CMA).
* Engaged in regular physical activity.
* Ankle considered healthy (no recent history of injury or instability).
* Verbal and written consent obtained.

Exclusion Criteria:

* History of ankle sprain, fracture, or surgery in the last 12 months.
* Musculoskeletal or neurological condition affecting walking or balance.
* Refusal to participate or withdrawal of consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Active military personnel in good health and performing operational duties (mainly infantrymen). Participants are recruited during periodic medical examinations at the 39th medical centre in Oberhoffen.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
Average Ankle-Go score in healthy military personnel | 6 months after the start of data collection
  Establish the mean value, standard deviation and reference intervals for the Ankle-Go score in a population of healthy military personnel, based on data collected during the complete test (physical tests and questionnaires). All these measurements correspond to a score (for example, for time in seconds, a patient performing exercise in 5 seconds, get a score of 2). All scores will be added together to obtain a single value considered as the final score.

CONTACTS AND LOCATIONS:
Locations (1):
- Cma05/Am039, Haguenau, France, France